CLINICAL TRIAL: NCT01565044
Title: Automatic Versus Intentional Movement Exercises to Enhance Arm Functions After Stroke
Acronym: AUTOTAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011.675
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Upper-limb Paresis
Keywords: Stroke; hemiplegia; automatic pilot; upper-limb rehabilitation
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- " AUTO " Group (Experimental)
  Interventions: Other: motor training
- " CONTROL " Group (Sham Comparator)
  Interventions: Other: motor training

INTERVENTIONS:
Other: motor training — Subject will perform prehension exercises on an automated table. After the initiation of the arm movement, the target to be grasped is programmed to move in order to stimulate automatic motricity.
  Arms: " AUTO " Group
Other: motor training — Subject will perform prehension exercises on an automated table. After the initiation of the arm movement, the target to be grasped will remain static in order to involve intentional motricity.
  Arms: " CONTROL " Group

SUMMARY:
Many patients retain upper-limb motor impairment following stroke. Most conventional rehabilitation techniques are aimed to improve motor intentional movement by repeated exercises. These techniques require attentional load and are responsible for significant fatigue that probably represents a limiting factor. Alternatively, the automatic control of action is now well documented. A rehabilitation method based on this principle could allow recovery of more natural movements.

Hypothesis: Stimulating automatic motricity improves upper-limb motor skills compared with a rehabilitation technique based on intentional movements.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be between the ages of 18-80 and must not be pregnant
* Patients volunteer to participate in the study, with a written informed consent signed
* Affiliation to a national health insurance program
* Hemiplegia after stroke
* Stroke onset >6 weeks and <4 years prior to study enrollment
* Patients able to perform the exercises on the automated table

Exclusion Criteria:

* Pregnancy
* Excessive pain in any joint of the paretic extremity (VAS>5)
* Coexistent major neurological or psychiatric disease as to decrease number of confounders
* Subjects with global aphasia and deficits of comprehension
* Any substantial decrease in alertness, language reception, or attention that might interfere with understanding instructions for motor testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer assessment (upper extremity) of motor recovery following stroke | 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during this follow-up session (Day 26).

SECONDARY OUTCOMES:
Fugl Meyer assessment (upper extremity) of motor recovery following stroke | immediately following the last day of the intervention (Day 12)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session
modified Ashworth scale | immediately following the last day of the intervention (Day 12) and 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session.
Visual Analog Pain Scale | immediately following the last day of the intervention (Day 12) and 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session.
Box and block test | immediately following the last day of the intervention (Day 12) and 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session
Frenchey Arm Test | immediately following the last day of the intervention (Day 12) and 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session.
Motor Activity Log (MAL | immediately following the last day of the intervention (Day 12) and 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session.
Functional independence scale (MIF) | immediately following the last day of the intervention (Day 12) and 2 weeks following the last day of the intervention (Day 26)
  we are looking for a change in scores between the baseline session score (Day 1), and those collected during each follow-up session

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Physique et de Réadaptation et Plateforme 'Mouvement et Handicap', Hôpital Henry Gabrielle, HCL, Saint-Genis-Laval, France